CLINICAL TRIAL: NCT01074437
Title: A Phase II, Randomized, Double-Blind Comparison of Corticosteroid and Corticosteroids With Propranolol Treatment of Infantile Hemangiomas (IH)
Brief Title: Corticosteroids With Placebo Versus Corticosteroids With Propranolol Treatment of Infantile Hemangiomas (IH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Jonathan Perkins, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12901
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-09

CONDITIONS: Hemangioma
MeSH Terms: conditions — Hemangioma | interventions — Prednisolone; Adrenal Cortex Hormones; Propranolol; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: Corticosteroid with Placebo (Other): Group A will receive oral, liquid Prednisolone, which is the standard corticosteroid that we use here at Seattle Children's, and oral liquid placebo. The dose of prednisolone that Group A will receive will be 1-2mg/kg/day for 7 days and then the dose will be slowly reduced and then stopped after 3 weeks. This is a standard dose for IH treatment. Gastric prophylaxis (Zantac) will be given to help prevent any stomach problems associated with prednisolone. This treatment will be given for two months, as is our standard practice.
  Interventions: Drug: Prednisolone (Corticosteroid); Drug: Placebo
- Group B: Corticosteroid with Propranolol (Other): Group B will receive oral liquid prednisolone, and oral propranolol. As in Group A, the dose of prednisolone will be 1-2mg/kg/day for 7 days and then the dose will be slowly reduced and then stopped after 3 weeks. Oral liquid propranolol will be dosed at 2 mg/kg/day, following initiation in the Cardiology Clinic. Gastric prophylaxis (Zantac) will be given to help prevent any stomach problems associated with prednisolone.
  Interventions: Drug: Prednisolone (Corticosteroid); Drug: Propranolol

INTERVENTIONS:
Drug: Prednisolone (Corticosteroid) — Oral liquid prednisolone. Dose: 1-2mg/kg/day for 7 days, and then dose will be slowly reduced and then stopped after 3 weeks.
  Other Names: Corticosteroids
Drug: Propranolol — Oral liquid propranolol will be dosed Oral liquid propranolol will be dosed at 2 mg/kg/day.
  Other Names: Propranolol hydrochloride (USP/EP) Oral Solution
  Arms: Group B: Corticosteroid with Propranolol
Drug: Placebo — Liquid placebo will be given during the two month treatment trial.
  Other Names: Inactive drug; Inactive substance; Inactive medicine
  Arms: Group A: Corticosteroid with Placebo

SUMMARY:
This is a prospective randomized, double-blind study to compare the clinical efficacy of infantile hemangioma treatment using propranolol with corticosteroids as compared to therapy with corticosteroids and placebo. We hypothesize that a two-month treatment period with propranolol plus corticosteroids is more effective at reducing infantile hemangioma size and vascularity when compared to corticosteroids used without propranolol for the same time period.

DETAILED DESCRIPTION:
Infantile hemangiomas (IH) are the most common head and neck pediatric tumors. Presence of these tumors can lead to complications of vision and airway compromise, bleeding and disfigurement. Medical treatment of these lesions has traditionally been focused on stopping new blood vessel growth with corticosteroids. Recent reports and our own experience have demonstrated that significant reduction in IH size and vascularity can also occur through the use of propranolol. Our initial experience with propranolol has demonstrated significant efficacy with fewer side effects than corticosteroids. Despite this experience, the standard of care for initial IH medical therapy remains corticosteroids.

This Trial is a direct comparison of traditional IH therapy with corticosteroids to newer therapy with propranolol and corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Age 0 to < 9months
* Patients with clinical, radiographic or histologic diagnosis of infantile hemangioma (IH) requiring medical treatment
* IH patients whose parents desire medical treatment for the IH
* Stable cardiac function

Exclusion Criteria:

* IH patients over 9 months of age.
* Hypersensitivity to propranolol
* Untreated heart failure: If the patient has heart failure associated with the hemangioma, propranolol would be initiated after anti-congestive therapy and under observation as an in-patient.
* Atrioventricular (AV) block
* Resting heart < 2 SD of normal*(below)
* Resting blood pressure < 2 SD of normal**(below)
* Wolff-Parkinson-White syndrome (WPW)
* History of unexplained syncope
* Bronchial asthma
* History of impaired renal or liver function
* Diabetes mellitus

Max Age: 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A Perkins, DO, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- [Background] Cushing SL, Boucek RJ, Manning SC, Sidbury R, Perkins JA. Initial experience with a multidisciplinary strategy for initiation of propranolol therapy for infantile hemangiomas. Otolaryngol Head Neck Surg. 2011 Jan;144(1):78-84. doi: 10.1177/0194599810390445. PMID 21493392
- [Background] Truong MT, Perkins JA, Messner AH, Chang KW. Propranolol for the treatment of airway hemangiomas: a case series and treatment algorithm. Int J Pediatr Otorhinolaryngol. 2010 Sep;74(9):1043-8. doi: 10.1016/j.ijporl.2010.06.001. Epub 2010 Jul 31. PMID 20674045

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A: Corticosteroid With Placebo | Group B: Corticosteroid With Propranolol
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Corticosteroid With Placebo | Group B: Corticosteroid With Propranolol | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 5 | 9
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.2 (0.1) | 0.2 (0.1) | 0.2 (0.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Compare Changes in IH Size and Vascularity for the Two Treatment Groups
Description: This outcome cannot be evaluated. Trial limited by lack of patient family to have randomization, which limited the number of participants and made the project nonviable.
Time Frame: 1, 2, and 6 months after treatment initiation
Population: This outcome cannot be evaluated. Trial limited by lack of patient family to have randomization, which limited the number of participants and made the project nonviable.
Arm/Group | Group A: Corticosteroid With Placebo | Group B: Corticosteroid With Propranolol
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Lesion Regression
Description: measure of change in lesion area or volume
Time Frame: 12 months
Population: Insufficient enrollment for data analysis to be meaningful.
Arm/Group | Group A: Corticosteroid With Placebo | Group B: Corticosteroid With Propranolol
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Determine Therapeutic Response of IH to Propranolol Among Patients Who Switch to Corticosteroids Plus Propranolol Therapy After Failing to Respond to Corticosteroids Alone.
Description: as for outcome 1
Time Frame: 1, 2, and 6 months after treatment initiation
Population: as for outcome 1
Arm/Group | Group A: Corticosteroid With Placebo | Group B: Corticosteroid With Propranolol
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Assess the Safety of Propranolol With Corticosteroids and Corticosteroids Alone in the Treatment of IH.
Description: as for outcome 1
Time Frame: 1, 2 and 6 months after treatment initiation
Population: as for outcome 1
Arm/Group | Group A: Corticosteroid With Placebo | Group B: Corticosteroid With Propranolol
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Demonstrate How Duplex Scanning to Assess Blood Vessel Density and Qualitative Color Ratings of Cutaneous Lesions From Photographs Can be Used to Measure and Quantify Changes in IH Size and Vascularity in a Clinically Relevant Manner.
Description: as for outcome 1
Time Frame: 1, 2 and 6 months after treatment initiation
Population: as for outcome 1
Arm/Group | Group A: Corticosteroid With Placebo | Group B: Corticosteroid With Propranolol
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group A: Corticosteroid With Placebo | Group B: Corticosteroid With Propranolol
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

LIMITATIONS AND CAVEATS:
Trial limited by lack of patient family to have randomization, which limited the number of participants and made the project nonviable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes